CLINICAL TRIAL: NCT01611532
Title: An Observational Study of the Role of Intra-abdominal Pressure Monitoring in Patients With Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Emma Aitken (Other)
Responsible Party: Sponsor-Investigator, Emma Aitken, Surgical Registrar, NHS Greater Glasgow and Clyde
Organization: NHS Greater Glasgow and Clyde (Other)
Other Study IDs: 11/WS/0040
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis; Intraabdominal pressure; Critical illness
MeSH Terms: conditions — Pancreatitis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute pancreatitis: All adult patients (>18y.o.) requiring admission for acute pancreatitis (amylase >3 times the upper limit of normal and typical symptoms of abdominal pain and vomiting)

SUMMARY:
Acute pancreatitis is a multi-system disease with an unpredictable clinical course and significant morbidity and mortality Approximately 20% of patients develop multi-organ failure requiring management within a critical care environment However much of the pathophysiology of the disease, particularly understanding why some patients develop life-threatening disease whilst others have a relatively benign course, remains unclear.

It well recognised that intra-abdominal hypertension (IAH) is a cause for organ dysfunction in critically ill patients and is associated with higher morbidity and mortality rates (Sugrue et al., 1999). Abdominal compartment syndrome (defined as an increase in intra-abdominal pressure (IAP) >20mmHg) is associated with new organ failure (Malbrain et al., 2006). The mechanisms believed to contribute to IAH in acute pancreatitis include increased capillary permeability, hypoalbuminaemia and volume overload ("third space losses"), producing retroperitoneal and visceral oedema (Dambrauskas et al., 2009).

Several small studies have recently described the link between intra-abdominal hypertension and adverse outcome in acute pancreatitis ( Dambrauskas et al., 2009; de Waele et al., 2005), however none of the authors appreciate the potential predictive value of there conclusions or the potential as a target for therapeutic intervention to alter the disease course.

This study aims to study the natural history of intra-abdominal pressures in acute pancreatitis and determine whether they truly do have a predictive value or whether they are simply another marker of organ failure in a multi-system disease with notoriously poor outcome.

DETAILED DESCRIPTION:
Acute pancreatitis is a multi-system disease with an unpredictable clinical course and significant morbidity and mortality (Wilmer, 2004). Approximately 20% of patients develop multi-organ failure requiring management within a critical care environment (Dambrauskas et al., 2009). However much of the pathophysiology of the disease, particularly understanding why some patients develop life-threatening disease whilst others have a relatively benign course, remains unclear.

Many predictive scales have resulted from attempts to predict which patients are likely to develop severe disease (Imrie, Ranson, APACHE-II etc.) (Barreto & Rodriguez, 2007). However none of these scoring systems actually correlate clinical findings with the pathophysiology of the disease process, making comprehension of the rationale for the prognostic value which these scales have been shown to have difficult. This has lead latterly to interest in measurement of intra-abdominal pressures (IAP) as a potential novel method to predict outcome in acute pancreatitis (Buter et al., 2002) since intra-abdominal hypertension can be explained by the disease processes in acute pancreatitis.

It well recognised that intra-abdominal hypertension (IAH) is a cause for organ dysfunction in critically ill patients and is associated with higher morbidity and mortality rates (Sugrue et al., 1999). Abdominal compartment syndrome (defined as an increase in IAP >20mmHg) is associated with new organ failure (Malbrain et al., 2006). The mechanisms believed to contribute to IAH in acute pancreatitis include increased capillary permeability, hypoalbuminaemia and volume overload ("third space losses"), producing retroperitoneal and visceral oedema (Dambrauskas et al., 2009).

Several small studies have recently described the link between intra-abdominal hypertension and adverse outcome in acute pancreatitis ( Dambrauskas et al., 2009; de Waele et al., 2005), however none of the authors appreciate the potential predictive value of there conclusions or the potential as a target for therapeutic intervention to alter the disease course.

This study aims to study the natural history of intra-abdominal pressures in acute pancreatitis and determine whether they truly do have a predictive value or whether they are simply another marker of organ failure in a multi-system disease with notoriously poor outcome.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >18y.o.
* Diagnosis of acute pancreatitis (defined as an amylase >3 times the upper limit of normal and typical symptoms)

Exclusion Criteria:

* Inability to provide informed consent
* Declines participation
* Uretheral catheterisation not required on clinical grounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with a diagnosis of acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
30 day mortality | 30 days

SECONDARY OUTCOMES:
Length of hospital stay | days
Length of HDU/ICU admission | days

CONTACTS AND LOCATIONS:
Locations (1):
- Monklands District General Hospital, Airdrie, Lanarkshire, United Kingdom